CLINICAL TRIAL: NCT00941200
Title: Pharmacogenetic DNA Bank
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: PG01/02/09
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood collection
  Interventions: Biological: Blood collection

INTERVENTIONS:
Biological: Blood collection

SUMMARY:
Aims of Research Proposal:

1. To build a DNA bank in association with a comprehensive database of treatment outcomes and toxicities of cancer patients.
2. To carry out genotyping of potential candidate genes in relation to specific anti-cancer agents and to correlate genotype with treatment outcomes and toxicities.

The investigators hypothesize that genetic variations between different individuals and ethnic groups may account for inter-individual and inter-ethnic differences in treatment response and toxicities to anti-cancer therapy. The understanding of the contribution of these genetic variations may help to individualize therapy to optimize treatment outcomes and reduce toxicities. Patients will be recruited from the National University Hospital Cancer Centre. Any individual aged 18 or above who has been diagnosed with cancer is eligible. 20 ml of blood will be collected from each subject for DNA extraction and pharmacogenetics analysis. At the time of recruitment, demographic characteristics, cancer history, and past and present cancer treatment history of the study subject will be collected. The patients' progress will be followed up periodically (approximately every 6 months) through the medical records, and subsequent cancer treatments, progression of cancer, and survival outcome will be updated. Follow-up will occur until death. Important treatment information that will be collected include the drug regimen, drug doses, intent of treatment, aematologic and non-haematologic toxicities, and hospitalization episodes that may be related to treatment. Known functional single nucleotide polymorphisms (SNPs) of drug metabolizing enzymes, transporters and targets of different anti-cancer agents will be characterized. More comprehensive genotyping will be carried out in 'outliers' who experience exceptional toxicity or biological response to identify novel functional SNPs using high throughput sequencing techniques. Correlation will be made between genotype and treatment-related outcomes (tumor response, progression-free survival) and toxicities. For selected patients, lymphoblastoid transformation will be carried out to maintain an infinite supply of DNA.

ELIGIBILITY:
Inclusion Criteria:

* Any cancer patient who is aged >=18 is eligible.

Exclusion Criteria:

* Cancer patients who are below age 18 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual who has been diagnosed with cancer is eligible.
Sampling Method: Non-Probability Sample
Enrollment: 5000
Dates: Start 2009-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, MRCP, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Wei X, McLeod HL, McMurrough J, Gonzalez FJ, Fernandez-Salguero P. Molecular basis of the human dihydropyrimidine dehydrogenase deficiency and 5-fluorouracil toxicity. J Clin Invest. 1996 Aug 1;98(3):610-5. doi: 10.1172/JCI118830. PMID 8698850
- [Background] Goetz MP, Knox SK, Suman VJ, Rae JM, Safgren SL, Ames MM, Visscher DW, Reynolds C, Couch FJ, Lingle WL, Weinshilboum RM, Fritcher EG, Nibbe AM, Desta Z, Nguyen A, Flockhart DA, Perez EA, Ingle JN. The impact of cytochrome P450 2D6 metabolism in women receiving adjuvant tamoxifen. Breast Cancer Res Treat. 2007 Jan;101(1):113-21. doi: 10.1007/s10549-006-9428-0. Epub 2006 Nov 18. PMID 17115111